CLINICAL TRIAL: NCT01234103
Title: Preventing Health Damaging Behaviors in Male and Female Army Recruits
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of continue funding
Sponsor: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cherrie B. Boyer, PhD, Professor of Pediatrics, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: W81XWH-04-1-0159
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Results first posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Sexually Transmitted Infection (STI) Prevention; Unintended Pregnancy Prevention; Sexual Risk Reduction; Alcohol and Other Substance Use Prevention; Intimate Partner Violence Prevention
Keywords: sexually transmitted infection; sexual risk; HIV; young adults; cognitive-behavioral intervention
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preventing sexual health risks (Experimental): The over goal is to prevent STIs, unintended pregnancies, and related behaviors including sexual risk, alcohol and other substance misuse
  Interventions: Behavioral: Preventing Helath Damaging Health Behaviors in Male and Female Army Recruits
- Improving nutrition, fitness and injury prevention (Other): The goals are: (1) maintain and improve nutrition and physical fitness through healthier lifestyle and food choices; (2) reduce the risk of sports or physical training injuries and learning how to treat injuries; and (3) Learn to recognize stress and the steps you can take to reduce stress
  Interventions: Behavioral: Preventing Helath Damaging Health Behaviors in Male and Female Army Recruits

INTERVENTIONS:
Behavioral: Preventing Helath Damaging Health Behaviors in Male and Female Army Recruits — Groups will be randomly assigned to the sexual/substance use prevention intervention or the comparative/control intervention focused on impro risk Involves 10 hours of didactic presentations, interactive group discussions, skills-building exercises, and topic specific videos to reduce participants' risk for and acquisition of STIs, unintended pregnancies and their associated sexual and substance use behaviors.

SUMMARY:
Health damaging (risk) behaviors of young military personnel are reflections of health problems facing all young people in the U.S. Military life presents opportunities and challenges that may both protect against and place young troops at risk for health damaging behaviors. Challenges for maintaining a healthy armed force include high rates of sexually transmitted infections (STIs), unintended pregnancies (UIPs), misuse of alcohol and other substances. The common thread through these negative health outcomes is volitional behavior. Such behaviors do not only result in illness or injury, but also negatively impact performance of military duties and threaten military readiness. Despite military leadership in setting standards and policies regarding professional behavior and universal health care for preventing and eliminating such negative health outcomes, many health problems remain. Building on our previous military research, we will evaluate the effectiveness a cognitive-behavioral, skills-building intervention to prevent and reduce young troops' risk for and acquisition of STIs and UIPs and will seek to reduce a number of their associated risk factors including, alcohol misuse, other substance use, and victimization due to IPV in male and female U.S. Army soldiers who are receiving Advance Individual Training (AIT) in Fort Jackson, SC.

DETAILED DESCRIPTION:
The primary hypotheses to be tested in this research are as follows. AIT soldiers participating in the experimental STI/UIP prevention intervention will: (a) have increased knowledge about the risk factors for and prevention of STIs, UIPs, alcohol and other substances, and intimate partner violence (IPV); (b) be more highly motivated to change risk behaviors associated with STIs and UIPs; (c) have higher levels of skills to prevent risk behaviors associated with STIs and UIPs and skills; (d) engage in more health promoting behaviors and fewer risk behaviors associated with STIs and UIPs, and (e) have fewer STIs and UIPs post-intervention compared with AIT solders who participate in a comparable control intervention focused on increasing healthy eating, maintaining physical fitness, and preventing fitness-related injuries.

The overall goal of this research is to evaluate the effectiveness a cognitive-behavioral skills-building intervention to prevent risk for and acquisition of STIs and UIPs and will seek to reduce a number of their associated risk factors including, alcohol misuse, other substance use, IPV in AIT soldiers. Specifically, we will evaluate whether AIT soldiers who participate in the experimental intervention entitled, Staying Safe and in Control: Increasing Knowledge and Building Skills to Prevent Sexually Transmitted Infections and Unintended Pregnancies will reduce their risk for and acquisition of STIs, UIPs and their associated sexual and substance use behaviors compared with AIT soldiers who undergo the control intervention entitled, Fit You: Practical Tools for Healthy Eating, Physical Fitness, and Injury Prevention. This intervention will focus primarily on promoting healthy eating, maintaining physical fitness, and preventing work-related and exercise injury.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be 18 years of age or older, will be fluent in English, and able to provide written, informed consent.

Exclusion Criteria:

* AIT soldiers under the age of 18 will be excluded since it will be difficult to obtain parental consent. We anticipate that this exclusion will be rare.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 933 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cherrie B Boyer, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Fort Jackson Advance Individual Training Units, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaydos CA, Howell MR, Pare B, Clark KL, Ellis DA, Hendrix RM, Gaydos JC, McKee KT Jr, Quinn TC. Chlamydia trachomatis infections in female military recruits. N Engl J Med. 1998 Sep 10;339(11):739-44. doi: 10.1056/NEJM199809103391105. PMID 9731090
- [Background] Boyer CB, Shafer MA, Moncada J, Schachter J, Shaffer RA, Brodine SK. Sociodemographic, behavioral, and clinical factors associated with STDs in a national sample of women entering the US military. ISSTDR: Sexually Transmitted Infections. 2001:241-246.
- [Background] Shafer MA, Moncada J, Boyer CB, Betsinger K, Flinn SD, Schachter J. Comparing first-void urine specimens, self-collected vaginal swabs, and endocervical specimens to detect Chlamydia trachomatis and Neisseria gonorrhoeae by a nucleic acid amplification test. J Clin Microbiol. 2003 Sep;41(9):4395-9. doi: 10.1128/JCM.41.9.4395-4399.2003. PMID 12958275
- [Background] Centers for Disease Control and Prevention. Sexually Transmitted Disease Surveillance 2000. Atlanta, GA: Division of Sexually Transmitted Diseases, National Center for HIV, STD and TB Prevention; 2001.
- [Background] Cecil JA, Howell MR, Tawes JJ, Gaydos JC, McKee KT Jr, Quinn TC, Gaydos CA. Features of Chlamydia trachomatis and Neisseria gonorrhoeae infection in male Army recruits. J Infect Dis. 2001 Nov 1;184(9):1216-9. doi: 10.1086/323662. Epub 2001 Sep 27. PMID 11598849
- [Background] Brodine SK, Shafer MA, Shaffer RA, Boyer CB, Putnam SD, Wignall FS, Thomas RJ, Bales B, Schachter J. Asymptomatic sexually transmitted disease prevalence in four military populations: application of DNA amplification assays for Chlamydia and gonorrhea screening. J Infect Dis. 1998 Oct;178(4):1202-4. doi: 10.1086/515685. PMID 9806061
- [Background] Shafer MA, Boyer CB, Shaffer RA, Schachter J, Ito SI, Brodine SK. Correlates of sexually transmitted diseases in a young male deployed military population. Mil Med. 2002 Jun;167(6):496-500. PMID 12099086
- [Background] Yen S, Shafer MA, Moncada J, Campbell CJ, Flinn SD, Boyer CB. Bacterial vaginosis in sexually experienced and non-sexually experienced young women entering the military. Obstet Gynecol. 2003 Nov;102(5 Pt 1):927-33. doi: 10.1016/s0029-7844(03)00858-5. PMID 14672465
- [Background] Howell MR, Gaydos JC, McKee KT Jr, Quinn TC, Gaydos CA. Control of Chlamydia trachomatis infections in female army recruits: cost-effective screening and treatment in training cohorts to prevent pelvic inflammatory disease. Sex Transm Dis. 1999 Oct;26(9):519-26. doi: 10.1097/00007435-199910000-00007. PMID 10534206
- [Background] Shafer MA, Pantell RH, Schachter J. Is the routine pelvic examination needed with the advent of urine-based screening for sexually transmitted diseases? Arch Pediatr Adolesc Med. 1999 Feb;153(2):119-25. doi: 10.1001/archpedi.153.2.119. PMID 9988241
- [Background] Magann EF, Nolan TE. Pregnancy outcome in an active-duty population. Obstet Gynecol. 1991 Sep;78(3 Pt 1):391-3. PMID 1876371
- [Background] McNeary AM, Lomenick TS. Military duty: risk factor for preterm labor? A review. Mil Med. 2000 Aug;165(8):612-5. PMID 10957855
- [Background] Clark JB, Holt VL, Miser F. Unintended pregnancy among female soldiers presenting for prenatal care at Madigan Army Medical Center. Mil Med. 1998 Jul;163(7):444-8. PMID 9695607
- [Background] United States Department of Health and Human Services. Alcohol research & health: highlights from the tenth special report to Congress, Health risks and benefits of alcohol consumption. Vol 24. Washington, DC: U.S. Government Printing Office; 2000.
- [Background] Bray RM, Fairbank JA, Marsden ME. Stress and substance use among military women and men. Am J Drug Alcohol Abuse. 1999 May;25(2):239-56. doi: 10.1081/ada-100101858. PMID 10395158
- [Background] Martin L. Personality characteristics that increase vulnerability to sexual harassment among U.S. Army soldiers. Mil Med. 2000 Oct;165(10):709-13. PMID 11050862
- [Background] Martin L, Rosen LN, Durand DB, Stretch RH, Knudson KH. Prevalence and timing of sexual assaults in a sample of male and female U.S. Army soldiers. Mil Med. 1998 Apr;163(4):213-6. PMID 9575764
- [Background] Sadler AG, Booth BM, Cook BL, Doebbeling BN. Factors associated with women's risk of rape in the military environment. Am J Ind Med. 2003 Mar;43(3):262-73. doi: 10.1002/ajim.10202. PMID 12594773
- [Background] Sadler AG, Booth BM, Nielson D, Doebbeling BN. Health-related consequences of physical and sexual violence: women in the military. Obstet Gynecol. 2000 Sep;96(3):473-80. doi: 10.1016/s0029-7844(00)00919-4. PMID 10960645
- [Background] Boyer CB, Barrett DC, Peterman TA, Bolan G. Sexually transmitted disease (STD) and HIV risk in heterosexual adults attending a public STD clinic: evaluation of a randomized controlled behavioral risk-reduction intervention trial. AIDS. 1997 Mar;11(3):359-67. doi: 10.1097/00002030-199703110-00014. PMID 9147428
- [Background] Boyer CB, Shafer MA, Tschann JM. Evaluation of a knowledge- and cognitive-behavioral skills-building intervention to prevent STDs and HIV infection in high school students. Adolescence. 1997 Spring;32(125):25-42. PMID 9105488
- [Background] The NIMH Multisite HIV Prevention Trial: reducing HIV sexual risk behavior. The National Institute of Mental Health (NIMH) Multisite HIV Prevention Trial Group. Science. 1998 Jun 19;280(5371):1889-94. doi: 10.1126/science.280.5371.1889. PMID 9632382
- [Background] Shain RN, Piper JM, Newton ER, Perdue ST, Ramos R, Champion JD, Guerra FA. A randomized, controlled trial of a behavioral intervention to prevent sexually transmitted disease among minority women. N Engl J Med. 1999 Jan 14;340(2):93-100. doi: 10.1056/NEJM199901143400203. PMID 9887160
- [Background] Boyer CB, Shafer MA, Shaffer RA, Brodine SK, Ito SI, Yniguez DL, Benas DM, Schachter J. Prevention of sexually transmitted diseases and HIV in young military men: evaluation of a cognitive-behavioral skills-building intervention. Sex Transm Dis. 2001 Jun;28(6):349-55. doi: 10.1097/00007435-200106000-00009. PMID 11403194
- [Background] Boyer CB, Shafer MA. Preventing STDs and unplanned pregnancies: a cognitive-behavioral intervention for young women entering the U.S. military. Journal of Adolescent Health. 2003;32(2):129.
- [Background] Jenkins RA, Jenkins PR, Nannis ED, McKee KT Jr, Temoshok LR. Correlates of human immunodeficiency virus infection risk behavior in male attendees of a clinic for sexually transmitted disease. Clin Infect Dis. 2000 Apr;30(4):723-9. doi: 10.1086/313744. PMID 10770735
- [Background] Williams JO, Bell NS, Amoroso PJ. Drinking and other risk taking behaviors of enlisted male soldiers in the US Army. Work. 2002;18(2):141-50. PMID 12441578
- [Background] Fisher JD, Fisher WA, Williams SS, Malloy TE. Empirical tests of an information-motivation-behavioral skills model of AIDS-preventive behavior with gay men and heterosexual university students. Health Psychol. 1994 May;13(3):238-50. doi: 10.1037//0278-6133.13.3.238. PMID 8055859
- [Background] Chernesky M, Jang D, Luinstra K, Chong S, Smieja M, Cai W, Hayhoe B, Portillo E, Macritchie C, Main C, Ewert R. High analytical sensitivity and low rates of inhibition may contribute to detection of Chlamydia trachomatis in significantly more women by the APTIMA Combo 2 assay. J Clin Microbiol. 2006 Feb;44(2):400-5. doi: 10.1128/JCM.44.2.400-405.2006. PMID 16455891
- [Background] Chernesky MA, Jang DE. APTIMA transcription-mediated amplification assays for Chlamydia trachomatis and Neisseria gonorrhoeae. Expert Rev Mol Diagn. 2006 Jul;6(4):519-25. doi: 10.1586/14737159.6.4.519. PMID 16824026
- [Background] Levett PN, Brandt K, Olenius K, Brown C, Montgomery K, Horsman GB. Evaluation of three automated nucleic acid amplification systems for detection of Chlamydia trachomatis and Neisseria gonorrhoeae in first-void urine specimens. J Clin Microbiol. 2008 Jun;46(6):2109-11. doi: 10.1128/JCM.00043-08. Epub 2008 Apr 9. PMID 18400919
- [Background] Moncada J, Schachter J, Hook EW 3rd, Ferrero D, Gaydos C, Quinn TC, Willis D, Weissfeld A, Martin DH. The effect of urine testing in evaluations of the sensitivity of the Gen-Probe Aptima Combo 2 assay on endocervical swabs for Chlamydia trachomatis and neisseria gonorrhoeae: the infected patient standard reduces sensitivity of single site evaluation. Sex Transm Dis. 2004 May;31(5):273-7. doi: 10.1097/01.olq.0000124611.73009.d5. PMID 15107628
- [Background] Masek BJ, Arora N, Quinn N, Aumakhan B, Holden J, Hardick A, Agreda P, Barnes M, Gaydos CA. Performance of three nucleic acid amplification tests for detection of Chlamydia trachomatis and Neisseria gonorrhoeae by use of self-collected vaginal swabs obtained via an Internet-based screening program. J Clin Microbiol. 2009 Jun;47(6):1663-7. doi: 10.1128/JCM.02387-08. Epub 2009 Apr 22. PMID 19386838
- [Background] Schachter J, Chernesky MA, Willis DE, Fine PM, Martin DH, Fuller D, Jordan JA, Janda W, Hook EW 3rd. Vaginal swabs are the specimens of choice when screening for Chlamydia trachomatis and Neisseria gonorrhoeae: results from a multicenter evaluation of the APTIMA assays for both infections. Sex Transm Dis. 2005 Dec;32(12):725-8. doi: 10.1097/01.olq.0000190092.59482.96. PMID 16314767
- [Background] Serlin M, Shafer MA, Tebb K, Gyamfi AA, Moncada J, Schachter J, Wibbelsman C. What sexually transmitted disease screening method does the adolescent prefer? Adolescents' attitudes toward first-void urine, self-collected vaginal swab, and pelvic examination. Arch Pediatr Adolesc Med. 2002 Jun;156(6):588-91. doi: 10.1001/archpedi.156.6.588. PMID 12038892
- [Background] Centers for Disease Control and Prevention; Workowski KA, Berman SM. Sexually transmitted diseases treatment guidelines, 2006. MMWR Recomm Rep. 2006 Aug 4;55(RR-11):1-94. PMID 16888612

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preventing Sexual Health Risks | Improving Nutrition, Fitness and Injury Prevention
Started | 542 | 391
Completed (Each was enrolled at baseline, completed all intervention sessions, but no follow-up sessions.) | 542 | 391
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preventing Sexual Health Risks | Improving Nutrition, Fitness and Injury Prevention | Total
Number analyzed (Participants) | 540 | 393 | 933
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.77 (3.121) | 20.77 (3.124) | 20.77 (3.121)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 56 | 124
  Male | 472 | 337 | 809
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 84 | 67 | 151
  Not Hispanic or Latino | 455 | 325 | 780
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian | 7 | 7 | 14
  Asian/Pacific Islander | 28 | 10 | 38
  African American/Black | 115 | 83 | 198
  Hispanic/Latino/a | 84 | 67 | 151
  Caucasian/White | 279 | 206 | 485
  Other/Mixed Race | 26 | 19 | 45
  Missing Data | 1 | 1 | 2
Marital Status [Count of Participants; unit: Participants]
  Single/Never Married | 460 | 337 | 797
  Married | 76 | 50 | 126
  Separated/Divorce | 3 | 6 | 9
  Missing | 1 | 0 | 1
5 or more drinks of alcohol on 1 occassion-past 3 months [Count of Participants; unit: Participants]
  No alcohol past 3 months | 366 | 246 | 612
  Never | 41 | 21 | 62
  Once/month or less | 59 | 63 | 122
  2-3 times/month | 26 | 32 | 58
  1 or more times/week | 44 | 27 | 71
  Missing | 4 | 4 | 8
Number of sex partners -ever [Mean (Standard Deviation); unit: sex partners] | 10.09 (26.300) | 8.39 (10.272) | 9.36 (20.967)
Number of pregnancies (males and females) [Count of Participants; unit: Participants]
  None | 397 | 293 | 690
  1 | 78 | 58 | 136
  2 | 37 | 23 | 60
  3-5 | 23 | 16 | 39
  Missing Data | 5 | 3 | 8
Number of pregnancies unintended [Count of Participants; unit: Participants]
  None | 428 | 317 | 745
  1 | 68 | 50 | 118
  2 | 26 | 14 | 40
  3-5 | 11 | 7 | 18
  Missing Data | 7 | 5 | 12
Sexually transmitted infection diagnosed-ever [Count of Participants; unit: Participants]
  None | 512 | 363 | 875
  1 | 23 | 15 | 38
  2 | 5 | 8 | 13
  3 | 0 | 2 | 2
  Missing Data | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Sexually Transmitted Infections and the Self-reported Numbers of Unintended Pregnancies
Time Frame: 6 to 9 months
Population: No data were collected from participants. Participants only attended intervention sessions.
Arm/Group | Preventing Sexual Health Risks | Improving Nutrition, Fitness and Injury Prevention
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Self-reported Behavioral Measures Related to STI/HIV Prevention
Time Frame: 6 to 9 months
Population: No data were collected from participants. Participants only attended intervention sessions.
Arm/Group | Preventing Sexual Health Risks | Improving Nutrition, Fitness and Injury Prevention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: This was a behavioral education intervention and adverse event data were collected after each intervention session.
Arm/Group | Preventing Sexual Health Risks | Improving Nutrition, Fitness and Injury Prevention
All-Cause Mortality (participants affected / at risk) | 0/540 | 0/393
Serious Adverse Events (participants affected / at risk) | 0/540 | 0/393
Other Adverse Events (participants affected / at risk) | 0/540 | 0/393

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No